CLINICAL TRIAL: NCT00724100
Title: A Phase 1, Dose Escalation Study of the Safety and Pharmacokinetics of ALB 109564(a) Administered Intravenously Every 3 Weeks to Subjects With Advanced Solid Tumors
Brief Title: A Trial of ALB 109564(a) in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Albany Molecular Research, Inc. (Industry)
Collaborators: Westat (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMRI-564-101
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2011-09

CONDITIONS: Cancer
Keywords: Malignancy; Solid tumor; Tubulin inhibitor
MeSH Terms: conditions — Neoplasms | interventions — ALB 109564a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ALB 109564(a) (12´-methylthiovinblastine dihydrochloride) — Starting dose is 1.2 mg/m2. Standard dose increase, in the absence of limiting toxicity, is 50%. Each dose of ALB 109564(a) will be administered by intravenous infusion once every 3 weeks (21-day cycle) over a period of time up to approximately 30 minutes. Number of cycles: Maximum of 12, until disease progression, or unacceptable toxicity develops. Greater than 12 cycles if disease has not progressed after 12 cycles, with Investigator's and Sponsor's approvals.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of ALB 109564(a), a novel tubulin inhibitor, and to assess safety, pharmacokinetics, and anti-tumor activity in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is the first clinical study of ALB 109564(a), a tubulin inhibitor, interfering with tubulin polymerization, primarily targeting microtubules that compose the mitotic spindle, resulting in metaphase arrest. The motivation for the development of ALB 109564(a) is to create a molecule that will provide greater anti-tumor activity than other licensed vinca alkaloids, without increasing the level of toxicity often associated with such therapies.

The objectives of the proposed study are: (1) to determine the safety and tolerability, including the maximum tolerated dose (MTD) and dose limiting toxicity (DLT), of ALB 109564(a) administered intravenously every 3 weeks to subjects with advanced, treatment-refractory solid tumors; (2) to evaluate the pharmacokinetics of ALB 109564(a); and (3) to document any observed anti-tumor activity.

The starting dose of 1.2 mg/m2 once every 3 weeks is expected to ensure a safe first-in-human dose and allow increases of 50% with the first several subject cohorts. The first cohort will enroll 3 subjects, and the subsequent 3-subject cohorts will proceed according to a modified Fibonacci scheme. The standard dose increase, in the absence of dose limiting toxicity, will be 50%. However, once 1 subject experiences a DLT, or 2 or more subjects within a cohort experience ≥ Grade 2 drug-related adverse events, all subsequent dose escalations will occur at approximately 25% increments. In the case that the dose escalation increment is decreased to 25% following 2 or more subjects with ≥ Grade 2 drug-related events, the increment can subsequently be reset at 50% if, in the 2 successive cohorts, no DLTs are observed, and no more than 1 subject per cohort experiences a ≥ Grade 2 drug-related AE. DLT and MTD determinations will be made according to the first treatment cycle (single dose plus 3-week follow-up). The MTD will be declared as the highest level at which none of the original 3 subjects or no more than 1 of the expanded 6-subject cohort experiences a DLT. At the MTD level, subjects will be enrolled into two parallel groups: Group A, those with solid tumor of unrestricted tumor type, and Group B, those with primary tumor type of soft tissue sarcoma. Up to a total of 24 subjects will be enrolled at the MTD.

Subjects who tolerate treatment will be eligible to continue receiving treatment to a maximum of 12 cycles on the same 3-week schedule per the Investigator's medical judgment. Subjects whose disease has not progressed after 12 cycles of treatment with ALB 109564(a) may continue receiving treatment on the same 3-week cycle, with the same protocol assessments, contingent upon the Investigator's judgment and the Sponsor's approval.

The actual enrollment of subjects will be determined by the safety experience and the number of dose-escalation cohorts required to achieve the MTD. The projected enrollment is approximately 60 subjects for a total study duration of approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age.
* Histologically or cytologically confirmed solid tumor that is metastatic or progressive and for whom no standard therapy holds curative potential.
* Evaluable disease, measurable by either imaging using Response Evaluation Criteria in Solid Tumors (RECIST) or tumor marker(s).
* ECOG Performance Status of ≤ 2.
* Life expectancy of > 12 weeks.
* Laboratory values:
* Absolute neutrophil count ≥ 1,500 cells/μL.
* Platelets ≥ 100,000 cells/μL.
* Total bilirubin ≤ 1.5 × ULN.
* AST (SGOT) ≤ 2.5 × ULN.
* ALT (SGPT) ≤ 2.5 × ULN.
* Serum creatinine ≤ 1.5 mg/dL, or a measured creatinine clearance of ≥ 50 mL/min.
* Subjects with primary liver cancer or hepatic metastasis are eligible, if the following criteria are met:
* Total bilirubin ≤ 1.5 mg/dL.
* AST (SGOT) and ALT (SGPT) ≤ 5 × ULN.
* Severe liver dysfunction (Child-Pugh Class C or uncompensated Class B with persistent encephalopathy, persistent ascites, prothrombin time > 1.5 × ULN) is not present.
* Ascites, if present, is managed with diuretic agents or repeated paracentesis (required no more frequently than once per month).
* Esophageal bleeding and varices, if present, have been sclerosed or banded, and no bleeding episodes have occurred during the prior 6 months.
* Subjects with asymptomatic treated brain metastasis (surgical resection or radiotherapy) are eligible, if neurologically stable and have been off steroids and anticonvulsants required for symptom control for at least 3 months before Cycle 1, Day 1.

Exclusion Criteria:

* Women who are pregnant or lactating or of child-bearing potential, but not using adequate contraception.
* Receipt of chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) before starting ALB 109564(a).
* Presence of acute or chronic adverse toxicity due to prior chemotherapy that has not resolved to ≤ Grade 1, as determined using the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0.
* Major surgery within 4 weeks before starting ALB 109564(a).
* Peripheral neuropathy of Grade ≥ 2 by CTCAE v3.0.
* Evidence of autonomic or other neuropathic syndromes, including chronic constipation.
* Confirmed diagnosis of HIV.
* Active, uncontrolled infection or systemic inflammatory disease.
* Active hepatitis B or C or other active liver disease (other than malignancy).
* Contraindication to a vinca alkaloid.
* Use of any investigational agent within 4 weeks of starting ALB 109564(a).
* Uncontrolled intercurrent illness that would jeopardize the subject's safety, interfere with the objectives of the protocol, or limit the subject's compliance with study requirements, as determined by the Investigator in consultation with the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose limiting toxicity. | Every treatment cycle

SECONDARY OUTCOMES:
Anti-tumor activity (objective tumor response, time to progression, duration of response) | Following every even-numbered cycle

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cho, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Geoffrey Shapiro, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute; Eunice L. Kwak, MD, PhD, Principal Investigator — Massachusetts General Hospital; Sridhar Mani, MD, Principal Investigator — Montefiore-Einstein Cancer Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Montefiore-Einstein Cancer Center, The Bronx, New York